CLINICAL TRIAL: NCT00106145
Title: A Phase I Study of MK0752, a Notch Inhibitor, in Patients With Metastatic or Locally Advanced Breast Cancer and Other Solid Tumors
Brief Title: A Notch Signalling Pathway Inhibitor for Patients With Advanced Breast Cancer (0752-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0752-014; 2005_008
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Breast Cancer; Other Solid Tumors
Keywords: Advanced Breast Cancer; Solid Tumors; Advanced Solid Tumors

ARMS (5):
- Part I - Arm 1 (Experimental)
  Interventions: Drug: Comparator: MK0752, Notch Inhibitor
- Part II - Arm 1 (Experimental)
  Interventions: Drug: Comparator: MK0752, Notch Inhibitor - 450 mg
- Part III - Arm 1 (Experimental)
  Interventions: Drug: Comparator: MK0752, Notch Inhibitor - 3 days on, 4 off
- Part IV - Arm 1 (Experimental)
  Interventions: Drug: Comparator: MK0752, Notch Inhibitor - 1 day on, 6 off
- Part V - Arm 1 (Experimental)
  Interventions: Drug: Comparator: MK0752, Notch Inhibitor - 3 days on, 4 off 350 mg

INTERVENTIONS:
Drug: Comparator: MK0752, Notch Inhibitor — Dose escalating beginning with rising dose levels of 300, 450, and 600 mg/day in a continuous dosing schedule.
  Arms: Part I - Arm 1
Drug: Comparator: MK0752, Notch Inhibitor - 450 mg — Dose 450 mg capsules daily for 28 day cycles.
  Arms: Part II - Arm 1
Drug: Comparator: MK0752, Notch Inhibitor - 3 days on, 4 off — Dose escalating in a repeating intermittent dosing schedule of 3 days on and 4 days off at rising dose levels of 450, 600, 800, 1000, 1200, and 1400 mg/day.
  Arms: Part III - Arm 1
Drug: Comparator: MK0752, Notch Inhibitor - 1 day on, 6 off — Dose escalating in a repeating intermittent dosing schedule of 1 day on/6 days off at rising dose levels of 600, 900, 1200, 1500, 1800, 2400, 3200 mg/day once weekly and then increase at 33% increments.
  Arms: Part IV - Arm 1
Drug: Comparator: MK0752, Notch Inhibitor - 3 days on, 4 off 350 mg — Dose 350 mg capsules daily intermittent 3 days on/4 days off dosing. THIS DOSING SCHEDULE IS NO LONGER UNDER INVESTIGATION
  Arms: Part V - Arm 1

SUMMARY:
An investigational study to determine the safety/tolerability, and efficacy of a notch signaling pathway inhibitor in patients with metastatic or locally advanced breast cancer and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Women or men greater than or equal to 18 years of age
* ECOG status less than or equal to 2 (a measurement to determine your ability to perform daily activities)
* In Parts I, III, and IV, patient must have a histologically confirmed, metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist. There is no limit on the number of prior treatment regimens
* In Part II, only breast cancer patients are eligible
* In Part V, only patients with Numb negative breast cancer (i.e., tumor shows Numb immunoreactivity in less than 10% of the neoplastic cells assessed) are eligible
* Patient has recovered from and is at least 2 weeks from previous antineoplastic therapy, including chemotherapy, biological therapy (including Herceptin), hormonal therapy, radiotherapy, or surgery

Exclusion Criteria:

* Patient has had an investigational treatment in the preceding 21 days
* Uncontrolled congestive heart failure or myocardial infarction (heart attack) within 3 months of study start
* History of hepatitis B or C or HIV
* Patient has the presence of clinically apparent central nervous system metastases or carcinomatous meningitis. Patients with CNS metastases who have completed a course of radiotherapy and are clinically stable in the judgment of the investigator are eligible
* Patients with "currently active" second malignancy, other than non-melanoma skin cancer, should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for prior malignancy and are considered by their physician to be at <30% risk of relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability; MTD will be established | Day 1 to Day 28

SECONDARY OUTCOMES:
Overall tumor/disease response will be evaluated using RECIST criteria, radiographic and clinical evaluations | radigraphic evaluation = every 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Krop I, Demuth T, Guthrie T, Wen PY, Mason WP, Chinnaiyan P, Butowski N, Groves MD, Kesari S, Freedman SJ, Blackman S, Watters J, Loboda A, Podtelezhnikov A, Lunceford J, Chen C, Giannotti M, Hing J, Beckman R, Lorusso P. Phase I pharmacologic and pharmacodynamic study of the gamma secretase (Notch) inhibitor MK-0752 in adult patients with advanced solid tumors. J Clin Oncol. 2012 Jul 1;30(19):2307-13. doi: 10.1200/JCO.2011.39.1540. Epub 2012 Apr 30. PMID 22547604